CLINICAL TRIAL: NCT04174976
Title: Morbidity of Abdominal Wall Hernia Reconstruction With Mesh: Study of Environmental Risk Factors in the Operating Room in the CHRU of Nancy- a Prospective Study
Brief Title: Environmental Risk Factors of Mesh Infection After Abdominal Wall Hernia Repair
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2019PI187
Record Dates: First submitted 2019-11-21; First posted 2019-11-22 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-10

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Wall hernia repair: All patients admitted for wall hernia repair with mesh between 28/12/2017 and 28/12/2020.
  .
  Interventions: Procedure: wall hernia repair

INTERVENTIONS:
Procedure: wall hernia repair — Wall hernia repair with mesh

SUMMARY:
Mesh infection is the main complication in abdominal hernia repair. In case of infection, a conservative management of mesh is not always possible. The removal of the mesh (occurring in 5.1% to 8% of wall hernia repair) increases the risk of recurrence and surgical morbidity.

Within our digestive surgery department (CHRU de Nancy), an infection rate of 10.7% (32 cases out of 298 patients with wall hernia repair) was observed between January 2016 and December 2018. This rate is higher than those usually described in the literature.

Several studies have identified predictors of mesh infection and explantation after abdominal wall hernia repair. The influence of the operating environment (temperature, hygrometry, pressure, number of people present, etc.) has, to our knowledge, never been studied.

If the risk of prosthesis infection is influenced by one or more of these extrinsic characteristics, it is possible to act on these practices to reduce this risk.

The main purpose of this study is to identify the characteristics specific to the intervention and the operating environment associated with mesh infection after abdominal wall hernia reconstruction

DETAILED DESCRIPTION:
It's a prospective, mono-centric study carried out on a cohort of patients followed in the digestive surgery department of the CHRU of Nancy

All patients who underwent a wall hernia repair between 28/12/2017 and 28/12/2020 in the digestive and general surgery department of the CHU of Nancy were included.

During the operative time, the nurses have to fill a survey with characteristics specific to the intervention and the operating environment.

Patients in this study have been followed for at least one year at the Nancy CHRU in order to be aware of the occurence of mesh infection and surgery for mesh explantation.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted for wall hernia repair with mesh between 28/12/2017 and 28/12/2020

Exclusion Criteria:

* Emergency surgery
* Laparoscopic
* Pregnancy
* Adults under legal guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients admitted for wall hernia repair with mesh between 28/12/2017 and 01/01/2021 (expected number of approximately 300 patients) for which follow-up data will be available during the first post-operative year
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-12-28 (Actual); Primary Completion 2021-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with surgical site infection | up to 1 year
  patient has at least one of the following:
  purulent drainage from the deep incision. a deep incision that spontaneously dehisces, or is deliberately opened or aspirated by a surgeon, physician* or physician designee AND organism(s) identified from the deep soft tissues of the incision by a culture or non-culture based microbiologic testing method which is performed for purposes of clinical diagnosis or treatment (for example, not Active Surveillance Culture/Testing (ASC/AST)) or culture or non-culture based microbiologic testing method is not performed. A culture or non-culture based test from the deep soft tissues of the incision that has a negative finding does not meet this criterion. AND patient has at least one of the following signs or symptoms: fever (>38°C); localized pain or tenderness.
  an abscess or other evidence of infection involving the deep incision that is detected on gross anatomical or histopathologic exam, or imaging test.

SECONDARY OUTCOMES:
Number of participants with surgery for mesh explantation | up to 1 year
  Surgery for mesh explantation

CONTACTS AND LOCATIONS:
Overall Officials: Estelle Vigneron, Principal Investigator — CHU NANCY
Locations (1):
- Estelle Vigneron, Nancy, France

IPD SHARING:
Plan to Share IPD: No